CLINICAL TRIAL: NCT00506181
Title: Phase 3 Study of Probiotics, to Provide a Legitimate Reason for the Administration of Probiotic Therapy in the Hospitalized Patient, Particularly in Patients on Antibiotic Therapy
Brief Title: Probiotics: is it Really That Good? Cost-Effectiveness of Treating the in-Patient
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: probiotics-HMO-CTIL
Record Dates: First submitted 2007-07-22; First posted 2007-07-25 (Estimated); Last update posted 2007-07-25 (Estimated); Status verified 2007-07

CONDITIONS: Diarrhea; Clostridium Difficile
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- X (Active Comparator): receiving probiotics
  Interventions: Drug: probiotic mixture
- Y (Placebo Comparator)
  Interventions: Drug: Placebo
- Z (No Intervention)

INTERVENTIONS:
Drug: probiotic mixture — "Jarro-Dophilus" probiotic mixture (4,400,000,000 bacteria in each capsule). One capsule X2/day.
  Arms: X
Drug: Placebo
  Arms: Y

SUMMARY:
Medical literature has dealt with various perspectives of probiotic therapy - prevention of antibiotic associated diarrhoea, Clostridium difficile, etc.

However, there have been no published results which can provide a basis for a generalized recommendation or discouragement of probiotic use among various groups of hospitalized patients.

The hypothesis is that the benefit in probiotic therapy in the admitted patient is by far larger than the actual cost of therapy. This assumption is probably true for all admitted patients and for patients on antibiotic therapy in particular.

DETAILED DESCRIPTION:
Probiotics are known as a food supplement available worldwide as an OTC drug, with minimal side effects. Probiotics have also been recommended as a food supplement to patients suffering of antibiotic side effects and to those suffering of IBD or IBS.

All patients admitted to Internal Medicine and the Medical Intensive Care Unit will be randomly divided in a double blind fashion into two groups. Group One will be provided with the probiotic mixture - one capsule, two times per day. Group Two will receive a placebo. Group Three will receive no therapy.

Objective parameters such as duration of hospital stay, mortality and diarrhea frequency will be recorded. In addition, the frequency of CDT as well as blood and urine cultures will be examined. Furthermore, subjective measures will be examined by use of a questionnaire to be filled by the patient and/or his/her family members, or by the treating nurse.

Later the data will be processed and analyzed to compare between all the study participants and between the subgroups of the study (i.e. patients on specific antibiotic therapies).

For each patient, the experiment will last throughout his/her entire hospital stay.

The study is to last for one year and until 120 patients have participated.

ELIGIBILITY:
Inclusion Criteria:

* All patients hospitalized in the Department of Internal Medicine for a minimum duration of 3 days.
* Age (all >18) and gender are to have no impact on the usage of the drug.

Exclusion Criteria:

* patients who do not agree to participate in the study
* patients on an NPO (nothing per os) order, if NPO includes medications
* patients who suffer of Celiac disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2007-07; Study Completion 2008-07 (Estimated)

PRIMARY OUTCOMES:
Reduction of AAD & CDT, and thus less hospitalization days and lower costs. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Elchanan Fried, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel, Jerusalem, Israel